CLINICAL TRIAL: NCT02619565
Title: Prognostic Value of Recurrent Mutations in a Prospective Cohort of Myelodysplasia and Secondary Acute Myeloid Leukemias
Brief Title: Prospective Study of Molecular Predictors of Survival in Myelodysplastic Syndromes
Acronym: MDS04
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Groupe Francophone des Myelodysplasies (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Institut Cochin (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOM09236 - P081246
Record Dates: First submitted 2015-04-20; First posted 2015-12-02 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic syndromes; mutations; overall survival; prognosis
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood samples if evolution of the disease (Other): blood samples at Day 0 and also if there is an evolution of the disease
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — blood samples at Day 0 and also if there is an evolution of the disease

SUMMARY:
This study aims at prospectively enrolling a cohort of 400 incident cases of myelodysplastic syndromes (MDS) at diagnosis, to evaluate the impact of recurrent mutations on overall survival and event-free survival, using next generation sequencing. Patients are affected by ineffective hematopoiesis and a propensity to leukemia in the elderly with a global incidence of 10/100,000/year.

DETAILED DESCRIPTION:
Myelodysplastic syndromes (MDS) are a heterogeneous group of stem cell disorders characterized by ineffective hematopoiesis with dysplasia and a propensity to acute myeloid leukemia. Patients are affected in the elderly with a global incidence of 10/100,000/year.

During the past 3 years, a significant progress has been made in the understanding of molecular pathogenesis through identification of mutations in epigenetic genes like TET2, ASXL1, EZH2, RUNX1, DNMT3A, IDH1/2, transcription factors, signalling molecules, cohesion and splicing regulators. Inactivating mutations targeting the hematopoietic stem cell may alter its gene expression pattern and could be an early mechanism of clonal selection. However, a single genetic alteration does not readily recapitulate the apoptotic and dysplastic phenotype. Several clones may co-exist, but their architecture is still unclear.

This study aims at prospectively enrolling a cohort of 350 incident cases at diagnosis, to identify evaluate the impact of recurrent mutations on overall survival and event-free survival, using next generation sequencing.

Considering the current knowledge, investigators propose to:

* perform whole exome sequencing to identify new mutations in a subset of 30 patients at diagnosis and in 10/30 samples at follow-up, and validate the recurrence of the new mutations in a training set.
* validate a high throughput technology for extensive genotyping to determine the mutational status of 54 target genes in the entire prospective cohort.
* analyze the frequency and impact on phenotype, OS and EFS of the most frequent mutations including SF3B1, SRSF2, ZRSR2, U2AF1, TET2, ASXL1, EZH2, IDH1/2, DNMT3A, NRAS, TP53, and RUNX1 and possibly of the newly discovered new mutations. Individual follow-up will be 36 months.

As ancillary studies, the evolution of mutation profiles after leukemic transformation in 10/30 MDS tested by WES, or after evaluation of the response to treatments in 100 MDS included in clinical trials of the "Groupe Francophone des Myélodysplasies" will be analyzed.

Understanding clonal architecture at diagnosis and after leukemic transformation is crucial for the knowledge of the pathophysiology of MDS. Better knowledge could help to adapt the therapeutic strategy. The study will help to delineate the pattern of genes which mutations with independent prognostic value modify the natural course of the disease. Then, investigators will apply for a grant to support a medico-economic evaluation of the molecular diagnosis in MDS.

ELIGIBILITY:
Inclusion Criteria:

Myelodysplastic syndromes, mixed myelodysplastic/myeloproliferative disorders or secondary acute myeloid leukemia at diagnosis:

* De novo MDS subtype according to the WHO classification: RCMD and RA with or without ring sideroblasts, RAEB 1, or MDS-U, RAEB 2, therapy-related MDS or sAML, MDS/MPD.
* IPSS
* Documented chromosome 5 and 7 abnormality (del(5q) or -5, del(7q) or -7) by FISH analysis, if possible AND
* ECOG performance status ≤ 2
* Age ≥ 18 years
* Life expectancy ≥ 3 months
* Adequate renal and liver function (transaminases serum levels ≤ 3N; calculated creatinine clearance > 40 ml/min)
* Signed informed consent prior to start of any study-specific procedures
* Ability to participate to a clinical trial and adhere to study procedures

Exclusion Criteria:

* Active serious infection not controlled by oral or intravenous antibiotics
* Treatment with any investigational antileukemic agent or chemotherapy at least 6 weeks prior to study entry and lack of full recovery from side effects due to prior therapy independent of when that therapy were given
* Rapidly progressive disease with compromised organ function judged to be life-threatening by the Investigator
* Pregnant or lactating female
* Known human immunodeficiency virus (HIV) infection
* Known active hepatitis B and/or C virus infection
* ECOG performance status > 2
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2010-04-12 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who survived event-free | 5 years
Number of surviving patients | 5 years

SECONDARY OUTCOMES:
Number of mutations on event-free survival in myelodysplastic syndromes | 5 years
  prevalence of TET2 mutation and other karyotypic abnormalities
Number of medullary blast and Hemoglobin, platelet and neutrophil polynuclear | 5 years
  to evaluate response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Fontenay, MD, PhD, Study Chair — Assistance publique-Hôpitaux de Paris and Paris Descartes University.
Locations (1):
- Assistance publique-Hôpitaux de Paris, Hôpital Cochin, Paris, France

REFERENCES:
- [Background] Damm F, Kosmider O, Gelsi-Boyer V, Renneville A, Carbuccia N, Hidalgo-Curtis C, Della Valle V, Couronne L, Scourzic L, Chesnais V, Guerci-Bresler A, Slama B, Beyne-Rauzy O, Schmidt-Tanguy A, Stamatoullas-Bastard A, Dreyfus F, Prebet T, de Botton S, Vey N, Morgan MA, Cross NC, Preudhomme C, Birnbaum D, Bernard OA, Fontenay M; Groupe Francophone des Myelodysplasies. Mutations affecting mRNA splicing define distinct clinical phenotypes and correlate with patient outcome in myelodysplastic syndromes. Blood. 2012 Apr 5;119(14):3211-8. doi: 10.1182/blood-2011-12-400994. Epub 2012 Feb 17. PMID 22343920
- [Background] Delhommeau F, Dupont S, Della Valle V, James C, Trannoy S, Masse A, Kosmider O, Le Couedic JP, Robert F, Alberdi A, Lecluse Y, Plo I, Dreyfus FJ, Marzac C, Casadevall N, Lacombe C, Romana SP, Dessen P, Soulier J, Viguie F, Fontenay M, Vainchenker W, Bernard OA. Mutation in TET2 in myeloid cancers. N Engl J Med. 2009 May 28;360(22):2289-301. doi: 10.1056/NEJMoa0810069. PMID 19474426
- [Background] Kosmider O, Gelsi-Boyer V, Cheok M, Grabar S, Della-Valle V, Picard F, Viguie F, Quesnel B, Beyne-Rauzy O, Solary E, Vey N, Hunault-Berger M, Fenaux P, Mansat-De Mas V, Delabesse E, Guardiola P, Lacombe C, Vainchenker W, Preudhomme C, Dreyfus F, Bernard OA, Birnbaum D, Fontenay M; Groupe Francophone des Myelodysplasies. TET2 mutation is an independent favorable prognostic factor in myelodysplastic syndromes (MDSs). Blood. 2009 Oct 8;114(15):3285-91. doi: 10.1182/blood-2009-04-215814. Epub 2009 Aug 7. PMID 19666869
- [Background] Kosmider O, Gelsi-Boyer V, Ciudad M, Racoeur C, Jooste V, Vey N, Quesnel B, Fenaux P, Bastie JN, Beyne-Rauzy O, Stamatoulas A, Dreyfus F, Ifrah N, de Botton S, Vainchenker W, Bernard OA, Birnbaum D, Fontenay M, Solary E; Groupe Francophone des Myelodysplasies. TET2 gene mutation is a frequent and adverse event in chronic myelomonocytic leukemia. Haematologica. 2009 Dec;94(12):1676-81. doi: 10.3324/haematol.2009.011205. Epub 2009 Oct 1. PMID 19797729
- [Background] Nibourel O, Kosmider O, Cheok M, Boissel N, Renneville A, Philippe N, Dombret H, Dreyfus F, Quesnel B, Geffroy S, Quentin S, Roche-Lestienne C, Cayuela JM, Roumier C, Fenaux P, Vainchenker W, Bernard OA, Soulier J, Fontenay M, Preudhomme C. Incidence and prognostic value of TET2 alterations in de novo acute myeloid leukemia achieving complete remission. Blood. 2010 Aug 19;116(7):1132-5. doi: 10.1182/blood-2009-07-234484. Epub 2010 May 20. PMID 20489055
- [Background] Itzykson R, Kosmider O, Cluzeau T, Mansat-De Mas V, Dreyfus F, Beyne-Rauzy O, Quesnel B, Vey N, Gelsi-Boyer V, Raynaud S, Preudhomme C, Ades L, Fenaux P, Fontenay M; Groupe Francophone des Myelodysplasies (GFM). Impact of TET2 mutations on response rate to azacitidine in myelodysplastic syndromes and low blast count acute myeloid leukemias. Leukemia. 2011 Jul;25(7):1147-52. doi: 10.1038/leu.2011.71. Epub 2011 Apr 15. PMID 21494260
- [Background] Kosmider O, Delabesse E, de Mas VM, Cornillet-Lefebvre P, Blanchet O, Delmer A, Recher C, Raynaud S, Bouscary D, Viguie F, Lacombe C, Bernard OA, Ifrah N, Dreyfus F, Fontenay M; GOELAMS Investigators. TET2 mutations in secondary acute myeloid leukemias: a French retrospective study. Haematologica. 2011 Jul;96(7):1059-63. doi: 10.3324/haematol.2011.040840. Epub 2011 Apr 20. PMID 21508122
- [Background] Quivoron C, Couronne L, Della Valle V, Lopez CK, Plo I, Wagner-Ballon O, Do Cruzeiro M, Delhommeau F, Arnulf B, Stern MH, Godley L, Opolon P, Tilly H, Solary E, Duffourd Y, Dessen P, Merle-Beral H, Nguyen-Khac F, Fontenay M, Vainchenker W, Bastard C, Mercher T, Bernard OA. TET2 inactivation results in pleiotropic hematopoietic abnormalities in mouse and is a recurrent event during human lymphomagenesis. Cancer Cell. 2011 Jul 12;20(1):25-38. doi: 10.1016/j.ccr.2011.06.003. Epub 2011 Jun 30. PMID 21723201
- [Background] Kosmider O, Gelsi-Boyer V, Slama L, Dreyfus F, Beyne-Rauzy O, Quesnel B, Hunault-Berger M, Slama B, Vey N, Lacombe C, Solary E, Birnbaum D, Bernard OA, Fontenay M. Mutations of IDH1 and IDH2 genes in early and accelerated phases of myelodysplastic syndromes and MDS/myeloproliferative neoplasms. Leukemia. 2010 May;24(5):1094-6. doi: 10.1038/leu.2010.52. Epub 2010 Apr 8. No abstract available. PMID 20376084
- [Background] Damm F, Thol F, Kosmider O, Kade S, Loffeld P, Dreyfus F, Stamatoullas-Bastard A, Tanguy-Schmidt A, Beyne-Rauzy O, de Botton S, Guerci-Bresler A, Gohring G, Schlegelberger B, Ganser A, Bernard OA, Fontenay M, Heuser M. SF3B1 mutations in myelodysplastic syndromes: clinical associations and prognostic implications. Leukemia. 2012 May;26(5):1137-40. doi: 10.1038/leu.2011.321. Epub 2011 Nov 8. No abstract available. PMID 22064355
- [Background] Frisan E, Vandekerckhove J, de Thonel A, Pierre-Eugene C, Sternberg A, Arlet JB, Floquet C, Gyan E, Kosmider O, Dreyfus F, Gabet AS, Courtois G, Vyas P, Ribeil JA, Zermati Y, Lacombe C, Mayeux P, Solary E, Garrido C, Hermine O, Fontenay M. Defective nuclear localization of Hsp70 is associated with dyserythropoiesis and GATA-1 cleavage in myelodysplastic syndromes. Blood. 2012 Feb 9;119(6):1532-42. doi: 10.1182/blood-2011-03-343475. Epub 2011 Dec 12. PMID 22160620
- [Background] Damm F, Chesnais V, Nagata Y, Yoshida K, Scourzic L, Okuno Y, Itzykson R, Sanada M, Shiraishi Y, Gelsi-Boyer V, Renneville A, Miyano S, Mori H, Shih LY, Park S, Dreyfus F, Guerci-Bresler A, Solary E, Rose C, Cheze S, Prebet T, Vey N, Legentil M, Duffourd Y, de Botton S, Preudhomme C, Birnbaum D, Bernard OA, Ogawa S, Fontenay M, Kosmider O. BCOR and BCORL1 mutations in myelodysplastic syndromes and related disorders. Blood. 2013 Oct 31;122(18):3169-77. doi: 10.1182/blood-2012-11-469619. Epub 2013 Sep 18. PMID 24047651
- [Background] Damm F, Fontenay M, Bernard OA. Point mutations in myelodysplastic syndromes. N Engl J Med. 2011 Sep 22;365(12):1154-5; author reply 155. doi: 10.1056/NEJMc1108665. No abstract available. PMID 21992131
- See also: Cancer research for personalized medicine is a consortium dedicated to integrative research against cancer at the Assistance Publique-Hôpitaux de Paris — http://www.carpem.fr